CLINICAL TRIAL: NCT03472989
Title: The Effectiveness of Radial Extracorporeal Shockwave Therapy (rESWT), Sham- rESWT, Standardised Exercise Program or Usual Care for Patients With Plantar Fasciopathy. Study Protocol for a Double-blind, Randomised Sham- Controlled Trial
Brief Title: Plantar Fasciopathy and the Effectiveness of Radial Extracorporeal Shockwave Therapy, Physical Training or Usual Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Marte Heide, MD, Medical doctor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/1325
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Plantar Fascitis
Keywords: plantar fasciopathy; plantar fasciitis; radial extracorporeal shock wave therapy; sham- radial extracorporeal shock wave therapy; high-load strength training; foot orthosis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the four intervention groups in parallell for the duration of the study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The patients who receive rESWT or sham-rESWT will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Radial extracorporeal shock wave (Active Comparator): Active shock wave treatment. All patients will get standardized information and custom made foot orthosis.
  Interventions: Device: Radial extracorporeal shock wave
- Sham-radial extracorporeal shock wave (Sham Comparator): Sham- shock wave treatment. All patients will get standardized information and custom made foot orthosis.
  Interventions: Device: Sham-radial extracorporeal shock wave
- Standardized high-load exercise program (Active Comparator): High-load exercise treatment. All patients will get standardized information and custom made foot orthosis.
  Interventions: Behavioral: Standardized high-load exercise program
- Usual care (Active Comparator): Only standardized information and custom made foot orthosis
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Device: Radial extracorporeal shock wave — Patients will receive treatment once a week for 3 weeks. Treatment will be administered by using the rESWT device named Swiss DolorClast (EMS). 2000 impulses are implied via the power hand piece to the area of max tenderness at the insertion of the plantar fascia, with a pressure of 1.5-3 bars depending on what the patient tolerates. The treatments will be given by a trained physiotherapist at our Department.
  Patients will also receive standardized information at baseline, and will get custom made foot orthosis.
  Arms: Radial extracorporeal shock wave
Device: Sham-radial extracorporeal shock wave — Patients will receive the same treatment as the patients in the group receiving real shock waves, but no real shock waves are conducted. The probe is similar in design, sound and shape.
  Patients will also receive standardized information at baseline, and will get custom made foot orthosis.
  Arms: Sham-radial extracorporeal shock wave
Behavioral: Standardized high-load exercise program — Patients will be instructed to do 2 exercises: "Unilateral heel raise" and "unilateral leg squat" three times a week for 12 weeks. The patients will have a total of 8 sessions supervised by a physiotherapist at our Department.
  Patients will also receive standardized information at baseline, and will get custom made foot orthosis.
  Arms: Standardized high-load exercise program
Behavioral: Usual care — Patients will get standardized information as in the other three intervention groups with information on pathogenesis, etiology and prognosis, and they will get custom made foot orthosis
  Arms: Usual care

SUMMARY:
The purpose of this study is to evaluate whether radial extracorporeal shockwave therapy (rESWT), sham- rESWT or standardised exercise program is more effective on change in heel pain than usual care in the treatment of plantar fasciopathy.

The null hypothesis is: There is no difference between rESWT, sham- rESWT or standardised exercise program on change in heel pain (primary outcome) and functioning (secondary outcomes) compared to usual care in the treatment of plantar fasciopathy at 6 months follow-up (and secondary outcomes at the 12 months follow-up).

Alternative hypothesis is:

H1: There is a difference between rESWT and usual care on change in heel pain (and secondary outcomes) at the 6 months follow-up (and secondary outcomes at the 12 months follow-up).

H2: There is a difference between sham-rESWT and usual care on change in heel pain (and secondary outcomes ) at 6 months follow-up (and secondary outcomes at the 12 months follow-up).

H3: There is a difference between standardized exercise program and usual care on change in heel pain (and secondary outcomes) at 6 months follow- up (and secondary outcomes at the 12 months follow-up).

DETAILED DESCRIPTION:
Plantar fasciopathy is a common cause of plantar heel pain, with reported lifetime prevalence up to 10%. The choice of best practice in these patients is debated. Two randomised studies reported that Radial Extracorporeal Shock Wave Therapy (rESWT) is effective, but a meta-analysis concluded that due to methological limitations the evidence is questioned. There are few studies reporting the effect on exercise programs with high-load strength training, despite widespread use. The usual care at our outpatient clinic is information on the pathogenesis, etiology and prognosis. We give advice on using proper footwear, including foot orthosis and to accept pain to a certain level during activity. To our knowledge there are no other previous trials comparing rESWT, sham-rESWT and exercises to usual care. This trial is designed in order to provide results important for future clinical practice.

The patients who give their informed consent will be randomised into one of the four Groups; rESWT, sham-rESWT, standardized exercise or usual care. A computer generation randomisation schedule with blocks of 8, in a 1:1 ratio, will be performed by an external statistician and electronically concealed. All the patients regardless of group allocation will receive standardized information (oral and written) on the condition and get custom made foot orthosis made by an orthopedic technician at Sophies Minde AS.

The patients are blinded for rESWT/sham-rESWT, whereas blinding of the exercise group and usual care group is not possible. To evaluate the blinding of the rESWT, the patients are asked after the last treatment whether they believe that they have received real rESWT, sham-rESWT or if they do not know.

The patients will have follow-up at 3 months, 6 months and 12 months. The main outcome is change in heel pain (NRS) during activity at 6 months. Patient characteristics, anthropometric data and the duration of symptoms in the different groups will be registered at baseline, and presented as mean values (SD) for continuous variables or numbers (%) for categorical data. Pain and function scores will be presented as mean (SD). In addition to the two- group comparisons with t-tests, we will perform longitudinal data analysis and perform a mixed model analysis to compare differences between groups at follow- up with adjustment for scores at baseline and present mean differences (95% confidence intervals).

We will perform analysis regarding secondary outcome as stated above. In addition we will apply multivariable logistic and linear regression analysis to identify predictive factors as demographics, clinical and ultrasound findings for primary and secondary outcomes. Model building will be done in a way that is appropriate for the given sample sizes, by restricting the number of potential predictive factors and considering shrinkage methods to stabilise predictions.

Participants in the exercise group not attending 6 of 8 sessions with the physiotherapist or not completing 30 of 36 exercise sessions (3 sessions per week, 12 weeks) are regarded as non- adherence. In the rESWT and sham- rESWT group, participants not attending 2 of 3 sessions are regarded as non- adherence. They will be included in the intention- to- treat analysis. There will also be a separate intention-to- treat analysis with only adherent patients.

There will be performed a study evaluating the validity, reliability and responsiveness on the Foot Functional Index Revised Short Form.

ELIGIBILITY:
Inclusion Criteria:

* Pain with duration > 3 months localized in the proximal insertion of the plantar fascia on the medial calcaneal tuberosity.

Only patients with reported pain NRS 3 or more at activity at baseline, will be included in the trial.

* Tenderness to palpation corresponding to the painful area.
* Be residents of Norway, understand oral and written Norwegian.

Exclusion Criteria:

* Treatment with radial extracorporeal shock wave therapy the last 3 months.
* Spondylarthropathy or rheumatoid arthritis.
* Plantar fibromatosis.
* Tarsal tunnel syndrome.
* Polyneuropathy.
* Previous surgery with remaining osteosynthesis material in the foot or ankle.
* Contraindications for shock wave therapy ( use of anticoagulant drugs, pregnancy, bleeding disorders, epilepsy or pacemaker)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) | 6 months
  Change in heel pain (during activity the last week ). Numeric rating scale is a patient reported pain intensity scale ranging from 0 (no pain) to 10 (worst possible pain).

SECONDARY OUTCOMES:
Foot Functional Index, revised, short Version (FFI-RS) | 6 and 12 months
  Change in Foot Health status. Consists of 34 questions.
RAND- 12 | 6 and 12 months
  Health related quality of life. 12 items.
Numeric rating scale (NRS) | 6 and 12 months
  Change in heel pain (in rest the last week). Numeric rating scale is a patient reported pain intensity scale ranging from 0 (no pain) to 10 (worst possible pain).
Numeric rating scale (NRS) | 12 months
  Change in heel pain (in activity the last week).Numeric rating scale is a patient reported pain intensity scale ranging from 0 (no pain) to 10 (worst possible pain).
Patient Global Impression Of Change Scale (PGIC) | 6 and 12 months
  7-point scale ranging from "very much improved" to "very much worse"

CONTACTS AND LOCATIONS:
Overall Officials: Aasne Fenne Hoksrud, MD, PhD, Study Director — Oslo University hospital, Department of Physical Medicine and Rehabilitation
Locations (1):
- Oslo University Hospital, Ullevål, Oslo, Norway

REFERENCES:
- [Background] Rompe JD. Plantar fasciopathy. Sports Med Arthrosc Rev. 2009 Jun;17(2):100-4. doi: 10.1097/JSA.0b013e3181a3d60e. PMID 19440137
- [Background] Sun J, Gao F, Wang Y, Sun W, Jiang B, Li Z. Extracorporeal shock wave therapy is effective in treating chronic plantar fasciitis: A meta-analysis of RCTs. Medicine (Baltimore). 2017 Apr;96(15):e6621. doi: 10.1097/MD.0000000000006621. PMID 28403111
- [Background] Rathleff MS, Molgaard CM, Fredberg U, Kaalund S, Andersen KB, Jensen TT, Aaskov S, Olesen JL. High-load strength training improves outcome in patients with plantar fasciitis: A randomized controlled trial with 12-month follow-up. Scand J Med Sci Sports. 2015 Jun;25(3):e292-300. doi: 10.1111/sms.12313. Epub 2014 Aug 21. PMID 25145882
- [Background] Landorf KB. Plantar heel pain and plantar fasciitis. BMJ Clin Evid. 2015 Nov 25;2015:1111. PMID 26609884
- [Background] Gill LH. Plantar Fasciitis: Diagnosis and Conservative Management. J Am Acad Orthop Surg. 1997 Mar;5(2):109-117. doi: 10.5435/00124635-199703000-00006. PMID 10797213
- [Background] Ibrahim MI, Donatelli RA, Schmitz C, Hellman MA, Buxbaum F. Chronic plantar fasciitis treated with two sessions of radial extracorporeal shock wave therapy. Foot Ankle Int. 2010 May;31(5):391-7. doi: 10.3113/FAI.2010.0391. PMID 20460065
- [Background] Gerdesmeyer L, Frey C, Vester J, Maier M, Weil L Jr, Weil L Sr, Russlies M, Stienstra J, Scurran B, Fedder K, Diehl P, Lohrer H, Henne M, Gollwitzer H. Radial extracorporeal shock wave therapy is safe and effective in the treatment of chronic recalcitrant plantar fasciitis: results of a confirmatory randomized placebo-controlled multicenter study. Am J Sports Med. 2008 Nov;36(11):2100-9. doi: 10.1177/0363546508324176. Epub 2008 Oct 1. PMID 18832341
- [Background] Riel H, Jensen MB, Olesen JL, Vicenzino B, Rathleff MS. Self-dosed and pre-determined progressive heavy-slow resistance training have similar effects in people with plantar fasciopathy: a randomised trial. J Physiother. 2019 Jul;65(3):144-151. doi: 10.1016/j.jphys.2019.05.011. Epub 2019 Jun 13. PMID 31204294
- [Background] Rasenberg N, Riel H, Rathleff MS, Bierma-Zeinstra SMA, van Middelkoop M. Efficacy of foot orthoses for the treatment of plantar heel pain: a systematic review and meta-analysis. Br J Sports Med. 2018 Aug;52(16):1040-1046. doi: 10.1136/bjsports-2017-097892. Epub 2018 Mar 19. PMID 29555795
- [Background] Whittaker GA, Munteanu SE, Menz HB, Tan JM, Rabusin CL, Landorf KB. Foot orthoses for plantar heel pain: a systematic review and meta-analysis. Br J Sports Med. 2018 Mar;52(5):322-328. doi: 10.1136/bjsports-2016-097355. Epub 2017 Sep 21. PMID 28935689
- [Background] Frisaldi E, Shaibani A, Benedetti F. Why We should Assess Patients' Expectations in Clinical Trials. Pain Ther. 2017 Jun;6(1):107-110. doi: 10.1007/s40122-017-0071-8. Epub 2017 May 5. PMID 28477082
- [Background] Budiman-Mak E, Conrad KJ, Mazza J, Stuck RM. A review of the foot function index and the foot function index - revised. J Foot Ankle Res. 2013 Feb 1;6(1):5. doi: 10.1186/1757-1146-6-5. PMID 23369667
- [Background] Johnson JA, Maddigan SL. Performance of the RAND-12 and SF-12 summary scores in type 2 diabetes. Qual Life Res. 2004 Mar;13(2):449-56. doi: 10.1023/B:QURE.0000018494.72748.cf. PMID 15085917
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Derived] Roe C, Heide M, Soberg HL, Brunborg C, Hoksrud AF, Myhre K, Brox JI, Mork M. One-Year Trajectory of Pain, Function, and Health-Related Quality of Life in Patients With Plantar Fasciopathy. J Foot Ankle Res. 2025 Sep;18(3):e70067. doi: 10.1002/jfa2.70067. PMID 40671207
- [Derived] Mork M, Soberg HL, Heide M, Hoksrud AF, Groven KS, Brunborg C, Roe C. Predictors for pain and functioning in patients with plantar fasciopathy one year after inclusion in a treatment trial in specialist care. BMC Musculoskelet Disord. 2024 Dec 20;25(1):1049. doi: 10.1186/s12891-024-08187-2. PMID 39702178
- [Derived] Heide M, Roe C, Mork M, Myhre K, Brunborg C, Brox JI, Hoksrud AF. Is radial extracorporeal shock wave therapy (rESWT), sham-rESWT or a standardised exercise programme in combination with advice plus customised foot orthoses more effective than advice plus customised foot orthoses alone in the treatment of plantar fasciopathy? A double-blind, randomised, sham-controlled trial. Br J Sports Med. 2024 Jul 31;58(16):910-918. doi: 10.1136/bjsports-2024-108139. PMID 38904119
- [Derived] Heide M, Mork M, Roe C, Brox JI, Fenne Hoksrud A. The effectiveness of radial extracorporeal shock wave therapy (rESWT), sham-rESWT, standardised exercise programme or usual care for patients with plantar fasciopathy: study protocol for a double-blind, randomised, sham-controlled trial. Trials. 2020 Jun 29;21(1):589. doi: 10.1186/s13063-020-04510-z. PMID 32600386

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT03472989/SAP_000.pdf